CLINICAL TRIAL: NCT05700045
Title: Effect of Dexmedetomidine Combined With Ropivacaine Transverse Abdominal Plane Block (TAP) on Opioid Dosage After Cesarean Section Under Multimodal Analgesia
Brief Title: TAP Using Dexmedetomidine and Ropivacaine for Cesarean Section Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY-20222263-F-1
Record Dates: First submitted 2022-12-26; First posted 2023-01-26 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2022-11

CONDITIONS: Multimodal Analgesia; Cesarean Section
Keywords: dexmedetomidine; transversus abdominis plane block
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine + ropivacaine (Experimental): each side dexmedetomidine 0.5ug/kg+0.25% ropivacaine 20ml TAP block
  Interventions: Drug: Dexmedetomidine
- ropivacaine (No Intervention): each side 0.25% ropivacaine 20ml TAP block

INTERVENTIONS:
Drug: Dexmedetomidine — each side dexmedetomidine 0.5ug/kg TAP block
  Arms: dexmedetomidine + ropivacaine

SUMMARY:
To evaluate the effect of dexmedetomidine as an adjuvant of ropivacaine in the TAP block on cesarean section parturients under multimodal analgesia, optimize the multimodal analgesia program for cesarean section, and guide perioperative analgesia managemen。This is a single center, double-blind, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 1) 37-42 weeks of gestation

  2) Plan cesarean section

  3) Receiving patient controlled intravenous analgesia

  4) Age>18 years

  5) ASA（American Society of Anesthesiologists) grade I-III

  6) Voluntary participation and informed consent

Exclusion Criteria:

* 1)The anesthesia method for cesarean section is general anesthesia or intraspinal anesthesia, and epidural administration is used

  2) Combined with other opioids during operation

  3) High risk pregnancy (multiple pregnancy, in vitro pregnancy, etc.) or pregnancy related complications (hypertension, preeclampsia, chorioamnionitis, etc.)

  4) Times of previous cesarean section ≥ 3

  5) BMI ≥ 50kg/m2 is not suitable for TAP block

  6) Allergies or contraindications to the drugs involved in the study

  7) Combined with operations other than tubal ligation and ovariectomy

  8) Severe renal function impairment (SCR>176 µ mol/L and/or blood urea nitrogen>17.9 mmol/L), severe liver function impairment (ALT and/or aspartate aminotransferase exceed 3 times the upper limit of normal value)

  9) Increased risk of coagulation dysfunction or bleeding (PLT<80 × 109/L or international normalized ratio> 1.5)

  10) History of chronic pain or opiate abuse

  11) Other clinical trials in the last three months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Consumption of hydromorphone | 48 hours after surgery
  Consumption of hydromorphone 48 hours after surgery

SECONDARY OUTCOMES:
Consumption of hydromorphone | 24 hours after surgery
  Consumption of hydromorphone 24 hours after surgery
First time to press bolus | 48 hours after surgery
  Time between end of surgery and first time to press bolus
Attempts of pressing bolus | 48 hours after surgery
  Attempts of pressing bolus at 4 hours, 12 hours, 24 hours and 48 hours after surgery respectively
Numeric Rating Scale | 48 hours after surgery
  Numeric rating scale sores at rest , ambulation and uterine contraction. Postoperative pain will be scored on a scale of 0 to 10 on the NRS, with nil (0) representing no pain and 10 representing the worst imaginable pain.
Postoperative satisfaction | 48 hours after surgery
  Self-planned satisfaction with postoperative analgesia 0 point: dissatisfied, persistent pain, unable to sleep;
  1. point: satisfied, slight pain, pain when breathing deeply or coughing;
  2. points: very satisfied, painless when breathing deeply or coughing, quiet to sleep
Postoperative Ramsay score | 48 hours after surgery
  It divides a patient's level of sedation into six categories ranging from severe agitation to deep coma. Level 1 sober: the patient is anxious, restless or irritable; Level 2 sober: the patient is cooperative, has good orientation or is quiet; Level 3 sober: the patient only responds to commands; Level 4 sleep: the patient responds quickly to light tapping between the eyebrows or strong sound stimulation; Grade 5 sleep: the patient is slow to respond to light tapping between the eyebrows or strong sound stimulation; Grade 6 sleep: the patient has no response to light tapping between the eyebrows or strong sound stimulation.

OTHER OUTCOMES:
Incidence of adverse events | 48 hours after surgery
  Incidence of adverse events after surgery, eg, pruritus, postoperative nausea and vomiting, dizziness, and respiratory depression
Incidence of rescue analgesia | 48 hours after surgery
  Parturient women with the NRS at rest>3 points or the NRS with movement>6 points will be given hydromorphone 0.3-0.5mg for rescue analgesia

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Fourth military medical university, Xijing Hospital, Xi'an, Shannxi
  - Huang Nie, Xi'an

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT05700045/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT05700045/ICF_001.pdf